CLINICAL TRIAL: NCT04983082
Title: Portsmouth Clinical Outcomes REsearch Database (CORE-D)- a Research Database of Routine Electronically Recorded Patient Data to Model Adverse Clinical Outcomes and Healthcare Resource Usage
Brief Title: Portsmouth CORE-D Routine Care Data Repository
Acronym: CORE-D
Status: Recruiting | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHU/2021/11
Record Dates: First submitted 2021-06-23; First posted 2021-07-30 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Adult Hospital Patients at Risk of Adverse Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
An integrated database of depersonalised routine hospital patient data consisting of demographic and disease attributes, physiological or laboratory measurements, care contacts and interventions along with associated clinical outcomes. The database is an essential resource for the development and testing of risk models and classification systems, modified as necessary for patient subgroups, which can then be introduced into clinical care to improve patient outcomes. It can also be used for large scale simulations to evaluate interventions.

DETAILED DESCRIPTION:
The aims and objectives of this database of depersonalised routinely collected hospital patient data are to:

* Conduct epidemiological and observational studies of acute hospital care.
* Develop and use algorithms and risk models to identify the deteriorating / sick adult so that interventions and enhanced care can be provided in a timelier manner with consequent resource and outcome improvements. This covers both the deteriorating inpatient at risk of adverse outcomes and people in the local community at risk of hospitalisation or in need of other health services.
* Retrospectively evaluate interventions e.g. impact of system-wide clinical pathway introduction
* Conduct simulations of clinical pathways

ELIGIBILITY:
Inclusion Criteria:

* Adult presenting at the acute hospital or receiving services from the hospital

Exclusion Criteria:

* Adults who have registered an opt out of research with National Health Service (NHS) Digital
* Adults who have contacted the hospital to ask that their records are not to be included in this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The research database will hold data on adults who are treated by Portsmouth Hospitals University National Health Service Trust (PHU), either as an outpatient, Accident and Emergency (A&E) attender, day case or inpatient or have investigations carried out by PHU services Adult patients are defined by the National Health Service (NHS) as individuals over 16 years old. Data on service contacts and use will only be included where the patient was more than 16 years old at that time. None of the data included in the Clinical Outcomes analyses are collected specifically for the purposes of research. All datasets are routinely collected clinical datasets, collected for clinical use and clinical audit.
Sampling Method: Probability Sample
Enrollment: 750000 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
In-hospital death | At 24 hours after an observation assessment or physiological measurement
  Death during hospital admission
In-hospital death | 30 days after admission
  Death during hospital admission
Unanticipated ICU admission | At 24 hours after an observation assessment or physiological measurement
  Unanticipated ICU admission during hospital stay
Unanticipated ICU admission | 30 days after admission
  Unanticipated ICU admission during hospital stay
Cardiac arrest | At 24 hours after an observation assessment or physiological measurement
  Cardiac arrest during hospital stay
Cardiac arrest | 30 days after admission
  Cardiac arrest during hospital stay

SECONDARY OUTCOMES:
Diagnosis of Corona Virus Disease (COVID) infection | 48 hours after presentation
  Diagnosis of COVID-19
Diagnosis of Corona Virus Disease (COVID) infection | At 48 hours after an observation assessment or physiological measurement
  Diagnosis of COVID-19
Detection of Acute Organ Dysfunction | 24 hours after presentation
  Detection of acute organ dysfunction as measured by components of the Sequential Organ Failure Assessment (SOFA) Score
Detection of Acute Organ Dysfunction | 48 hours after presentation
  Detection of acute organ dysfunction as measured by components of the Sequential Organ Failure Assessment (SOFA) Score
Detection of Acute Organ Dysfunction | 72 hours after presentation
  Detection of acute organ dysfunction as measured by components of the Sequential Organ Failure Assessment (SOFA) Score
Detection of Acute Organ Dysfunction | 1 week after presentation
  Detection of acute organ dysfunction as measured by components of the Sequential Organ Failure Assessment (SOFA) Score
Detection of Acute Organ Dysfunction | 30 days after presentation
  Detection of acute organ dysfunction as measured by components of the Sequential Organ Failure Assessment (SOFA) Score

CONTACTS AND LOCATIONS:
Overall Officials: Paul E Schmidt, MRCP, Principal Investigator — Portsmouth Hospitals University NHS Trust
Locations (1):
- Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Bona fides United Kingdom (UK) researchers can make requests for access. They will be asked to detail their proposal in standard form which will be assessed by a Data Access Committee. Data will only be made available in a fully anonymous form and will be subject to a data sharing agreement.